CLINICAL TRIAL: NCT04405570
Title: A Phase IIa Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety, Tolerability and Efficacy of EIDD-2801 to Eliminate SARS-CoV-2RNA Detection in Persons With COVID-19
Brief Title: Safety, Tolerability and Efficacy of Molnupiravir (EIDD-2801) to Eliminate Infectious Virus Detection in Persons With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ridgeback Biotherapeutics, LP (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EIDD-2801-2003
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Results first posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: SARS-CoV-2 Infection, COVID-19
MeSH Terms: conditions — COVID-19 | interventions — molnupiravir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Molnupiravir 200 mg (Experimental): Molnupiravir 200 mg, twice daily (BID) for 5 days
  Interventions: Drug: Molnupiravir 200 mg
- Molnupiravir 400 mg (Experimental): Molnupiravir 400 mg, twice daily (BID) for 5 days
  Interventions: Drug: Molnupiravir 400 mg
- Molnupiravir 800 mg (Experimental): Molnupiravir 800 mg, twice daily (BID) for 5 days
  Interventions: Drug: Molnupiravir 800 mg
- Placebo (PBO) twice daily (BID) for 5 days (Placebo Comparator)
  Interventions: Drug: Placebo (PBO)

INTERVENTIONS:
Drug: Molnupiravir 200 mg — Oral capsule of molnupiravir
  Arms: Molnupiravir 200 mg
Drug: Molnupiravir 400 mg — Oral capsule of molnupiravir
  Arms: Molnupiravir 400 mg
Drug: Molnupiravir 800 mg — Oral capsule of molnupiravir
  Arms: Molnupiravir 800 mg
Drug: Placebo (PBO) — placebo oral capsule
  Arms: Placebo (PBO) twice daily (BID) for 5 days

SUMMARY:
This was a phase IIa, double-blind, placebo-controlled, randomized trial, designed to compare the safety, tolerability, and antiviral activity of EIDD-2801 (molnupiravir) versus placebo as measured by SARS-CoV-2 viral RNA detection in symptomatic adult outpatients with COVID-19.

DETAILED DESCRIPTION:
This was a phase IIa, double-blind, placebo-controlled, randomized trial, designed to compare the safety, tolerability, and antiviral activity of molnupiravir versus placebo as measured by SARS-CoV-2 viral RNA detection in symptomatic adult outpatients with COVID-19. The study was a multicenter trial that was conducted in the United States.

In this study, 204 participants were randomized and 202 received molnupiravir or placebo orally twice a day (BID) for 5 days. The study enrolled participants in 5 parts with each part evaluating molnupiravir doses of either 200 mg BID, 400 mg BID, or 800 mg BID. Doses were chosen based on emerging virology and safety data from this and ongoing studies. New dose groups were started after the selected dose had been studied for safety in a Phase 1 study.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent prior to initiation of any study procedures.
2. ≥18 years of age at Screening.
3. Study treatment is expected to begin within ≤168 hours from first symptom onset.
4. Ability to swallow pills.
5. Documentation of confirmed active SARS-CoV-2 infection, as determined by a molecular or non-molecular ("rapid") test conducted at any clinic or laboratory that had a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent from a sample collected ≤96 hours prior to study entry.
6. Was experiencing at least one of the following SARS-CoV-2 infection symptoms at the time of enrollment: fever (could be subjective including feeling feverish or having chills) OR signs/symptoms of respiratory illness (including but not limited to upper respiratory congestion, loss of sense of smell or taste, sore throat OR lower respiratory illness - cough, shortness of breath).
7. Agreed to not participate in another interventional clinical trial for the treatment of SARS-CoV-2 during the study period (28 days) unless hospitalized.
8. Agreed to not obtain investigational medications outside of the molnupiravir study.
9. Agreed to the sampling detailed in the schedule of evaluations and to comply with study requirements including contraception requirements.
10. A female participant was eligible to participate if she was not pregnant or breastfeeding and at least one of the following conditions applied:

    * Was not a woman of childbearing potential (WOCBP) OR
    * Was a WOCBP and using a contraceptive method that is highly effective (a low user dependency method OR a user-dependent method in combination with a barrier method), or was abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis), as described in Appendix 2 of the study protocol during the intervention period and for at least 50 days after the last dose of study intervention. The investigator evaluated the potential for contraceptive method failure (ie, noncompliance, recently initiated) in relationship to the first dose of study intervention.
    * A WOCBP must have had a negative highly sensitive pregnancy test (serum or urine) within 24 hours before the first dose of study intervention.
    * Additional requirements for pregnancy testing during and after study intervention were provided in the study protocol.
    * The investigator was responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
    * Contraceptive use by women was to be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
    * Given the elevated risk of venous thrombotic events in patients hospitalized with COVID-19 (Benson et al, 2020; Spratt et al, 2020), estrogen-containing contraceptives could not be started to fulfill the contraceptive requirement of this study at any time during participant's participation. If contraceptives were interrupted as standard of care management of COVID-19 patients and resumed at a later time point, such as at hospital discharge, then abstinence was practiced for the defined period of back-up contraception per the contraceptive product labeling. After this period, contraceptive use had to adhere to the guidance in Appendix 2 of the study protocol.
11. Male participants were eligible to participate if they agreed to the following during the intervention period and for at least 100 days after the last dose of study intervention:

    * Refrained from donating sperm

PLUS either:

* Were abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agreed to remain abstinent.

OR

* Had to agree to use contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause [Appendix 2 of the study protocol]) as detailed below:

  * Agreed to use a male condom plus partner use of an additional contraceptive method when having penile-vaginal intercourse with a WOCBP who was not pregnant. Note: Men with a pregnant or breastfeeding partner had to agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile-vaginal penetration.
  * Contraceptive use by men was to be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

1. Need for hospitalization or immediate medical attention in the clinical opinion of the study investigator.
2. Hemoglobin <10 g/dL in men and <9 g/dL in women.
3. Platelet count <100,000/ µL or received a platelet transfusion within 5 days prior to enrollment.
4. Was on dialysis or has an estimated glomerular filtration rate <30 mL/min/1.73 m^2
5. Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >3x upper limit normal (ULN).
6. History of or current hospitalization for COVID-19. Note: Individuals hospitalized and then discharged, even if only hospitalized for 1 day, were excluded.
7. History of kidney disease as evidenced by estimated creatinine clearance value <30 mL/min.
8. History of significant liver disease in the opinion of the site investigator or active hepatitis B or active hepatitis C. Human immunodeficiency virus (HIV) that is advanced (CD4<200/mm^3) and/or on treatment with nucleos(t)ide analogues.
9. Use of therapeutic interventions with possible anti-SARS-CoV-2 activity within 30 days prior to study entry, (e.g., remdesivir, lopinavir/ritonavir fixed dose combination, ribavirin, chloroquine, hydroxychloroquine, and convalescent plasma), or participation in a clinical trial involving any of these drugs whether for treatment or prophylaxis.
10. Receipt of a SARS-CoV-2 vaccination prior to study entry.
11. Known allergy/sensitivity or any hypersensitivity to components of molnupiravir, or its formulation.
12. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
13. History of recent (within the past 3 months) hemorrhagic cerebrovascular accident) or major bleed.
14. Presence of a condition, that in the opinion of the investigator, would place the subject at increased risk from study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2021-02-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Valley Clinical Trials, Inc., Northridge, California
  - FOMAT Medical Research, Oxnard, California
  - Southern California Emergency Medicine, Yucaipa, California
  - Indago Research and Health Center, Inc., Hialeah, Florida
  - NOLA Research Works, LLC, New Orleans, Louisiana
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Care United Research, LLC, Forney, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Mollan KR, Eron JJ, Krajewski TJ, Painter W, Duke ER, Morse CG, Goecker EA, Premkumar L, Wolfe CR, Szewczyk LJ, Alabanza PL, Loftis AJ, Degli-Angeli EJ, Brown AJ, Dragavon JA, Won JJ, Keys J, Hudgens MG, Fang L, Wohl DA, Cohen MS, Baric RS, Coombs RW, Sheahan TP, Fischer WA. Infectious Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Virus in Symptomatic Coronavirus Disease 2019 (COVID-19) Outpatients: Host, Disease, and Viral Correlates. Clin Infect Dis. 2022 Aug 24;75(1):e1028-e1036. doi: 10.1093/cid/ciab968. PMID 35022711
- [Derived] Fischer W, Eron JJ, Holman W, Cohen MS, Fang L, Szewczyk LJ, Sheahan TP, Baric R, Mollan KR, Wolfe CR, Duke ER, Azizad MM, Borroto-Esoda K, Wohl DA, Loftis AJ, Alabanza P, Lipansky F, Painter WP. Molnupiravir, an Oral Antiviral Treatment for COVID-19. medRxiv [Preprint]. 2021 Jun 17:2021.06.17.21258639. doi: 10.1101/2021.06.17.21258639. PMID 34159342
- [Derived] Mollan KR, Eron JJ, Krajewski TJ, Painter W, Duke ER, Morse CG, Goecker EA, Premkumar L, Wolfe CR, Szewczyk LJ, Alabanza PL, Loftis AJ, Degli-Angeli EJ, Brown AJ, Dragavon JA, Won JJ, Keys J, Hudgens MG, Fang L, Wohl DA, Cohen MS, Baric RS, Coombs RW, Sheahan TP, Fischer WA 2nd. Infectious SARS-CoV-2 Virus in Symptomatic COVID-19 Outpatients: Host, Disease, and Viral Correlates. medRxiv [Preprint]. 2021 Jun 25:2021.05.28.21258011. doi: 10.1101/2021.05.28.21258011. PMID 34100024
- [Derived] Cox RM, Wolf JD, Plemper RK. Therapeutically administered ribonucleoside analogue MK-4482/EIDD-2801 blocks SARS-CoV-2 transmission in ferrets. Nat Microbiol. 2021 Jan;6(1):11-18. doi: 10.1038/s41564-020-00835-2. Epub 2020 Dec 3. PMID 33273742
- See also: Benson et al, 2020. Society of Family Planning interim clinical recommendations — https://doi.org/10.46621/UYGR2287

RESULTS

PARTICIPANT FLOW:
Groups:
- Molnupiravir 200 mg; Molnupiravir 400 mg; Molnupiravir 800 mg: molnupiravir twice daily (BID) for 5 days
- Placebo: Placebo twice daily (BID) for 5 days
Period: Overall Study
Arm/Group | Molnupiravir 200 mg | Molnupiravir 400 mg | Molnupiravir 800 mg | Placebo
Started | 23 | 64 | 55 | 62
Number of Subjects Randomized Not Dosed | 0 | 2 | 0 | 0
Number of Subjects in the Safety Population | 23 | 62 | 55 | 62
Number of Subjects in the mITT Population | 23 | 61 | 53 | 61
Completed | 23 | 59 | 52 | 61
Not Completed | 0 | 5 | 3 | 1
Not completed — Adverse Event | 0 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Randomized not dosed | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Molnupiravir 200 mg | Molnupiravir 400 mg | Molnupiravir 800 mg | Placebo | Total
Number analyzed (Participants) | 23 | 62 | 55 | 62 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (15.34) | 42.4 (14.88) | 42.2 (14.36) | 39.7 (14.10) | 40.8 (14.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 32 | 27 | 34 | 104
  Male | 12 | 30 | 28 | 28 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 23 | 33 | 23 | 86
  Not Hispanic or Latino | 16 | 39 | 21 | 39 | 115
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 1 | 2 | 6
  Black or African American | 3 | 3 | 3 | 2 | 11
  White | 17 | 56 | 49 | 54 | 176
  Other | 2 | 0 | 2 | 1 | 5
  Multiple | 0 | 1 | 0 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Until First Non-detectable SARS-CoV-2 in Nasopharyngeal (NP) Swabs
Description: The number of participants until first non-detectable SARS-CoV-2 in nasopharyngeal (NP) swabs will be estimated for each randomized arm (drug versus placebo), using Kaplan-Meier methods with a corresponding log-rank test.
  Non detectable defined as "a viral load below the limit of quantification
Time Frame: 28 days
Population: mITT - modified Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Molnupiravir 200 mg | Molnupiravir 400 mg | Molnupiravir 800 mg | Placebo
Number analyzed (Participants) | 23 | 61 | 53 | 61
Participants
  Number (%) with response | 21 | 48 | 49 | 49
  Number (%) censored | 2 | 13 | 4 | 12
Statistical Analysis 1: Comparison: Molnupiravir 200 mg; Test type: Superiority; p = 0.5551, Log Rank
Statistical Analysis 2: Comparison: Molnupiravir 400 mg; Test type: Superiority; p = 0.7270, Log Rank
Statistical Analysis 3: Comparison: Molnupiravir 800 mg; Test type: Superiority; p = 0.0128, Log Rank

2. Primary Outcome: Time to Clearance of SARS-CoV-2 in Nasopharyngeal Swabs
Description: The distribution of days until first non-detectable SARS-CoV-2 in nasopharyngeal (NP) swabs will be estimated for each randomized arm (drug versus placebo), using Kaplan-Meier methods with a corresponding log-rank test.
  Non detectable defined as "a viral load below the limit of quantification
Time Frame: 28 days
Population: mITT - modified Intent to Treat Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Molnupiravir 200 mg | Molnupiravir 400 mg | Molnupiravir 800 mg | Placebo
Number analyzed (Participants) | 23 | 61 | 53 | 61
Days | 22.0 [15.0 to 28.0] | 27.0 [15.0 to 28.0] | 14.0 [13.0 to 14.0] | 15.0 [15.0 to 27.0]

3. Primary Outcome: Number of Participants With Adverse Events (AEs) Grade 3 or Higher or Leading to Discontinuation of Study Treatment
Description: 1) any AEs leading to early discontinuation of blinded treatment (active or placebo), 2) study drug-related discontinuation of treatment, 3) new grade 3 or higher AEs (not already present at baseline), and 4) study drug-related new grade 3 or higher AEs.
Time Frame: 28 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Molnupiravir 200 mg | Molnupiravir 400 mg | Molnupiravir 800 mg | Placebo
Number analyzed (Participants) | 23 | 62 | 55 | 62
Participants
  AEs leading to early discontinuation of blinded treatment (active or placebo) | 0 | 1 | 1 | 1
  AEs leading to study drug-related discontinuation of treatment | 0 | 0 | 0 | 0
  new grade 3 or higher AEs (not already present at baseline) | 1 | 2 | 4 | 5
  study drug-related new grade 3 or higher AEs | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Any Adverse Events (AEs), Grade 2 or Higher
Description: Measure the safety and tolerability of EIDD-2801 by estimating the occurrence of Grade 2 or higher AE and drug related AEs.
Time Frame: 28 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Molnupiravir 200 mg; Molnupiravir 400 mg; Molnupiravir 800 mg: EIDD-2801 twice daily (BID) for 5 days
Arm/Group | Molnupiravir 200 mg | Molnupiravir 400 mg | Molnupiravir 800 mg | Placebo
Number analyzed (Participants) | 23 | 62 | 55 | 62
Participants | 5 | 7 | 6 | 9

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Molnupiravir 200 mg | Molnupiravir 400 mg | Molnupiravir 800 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/62 | 0/55 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/23 | 2/62 | 1/55 | 1/62
Other Adverse Events (participants affected / at risk) | 4/23 | 2/62 | 1/55 | 4/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Molnupiravir 200 mg (N=23) | Molnupiravir 400 mg (N=62) | Molnupiravir 800 mg (N=55) | Placebo (N=62)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Molnupiravir 200 mg (N=23) | Molnupiravir 400 mg (N=62) | Molnupiravir 800 mg (N=55) | Placebo (N=62)
Dizziness (Nervous system disorders) | 2 (2) | 1 (3) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is requested to obtain written consent from the Sponsor before anything relating to the study can be published.

DOCUMENTS (2):
  • Study Protocol (2020-11-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT04405570/Prot_003.pdf
  • Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT04405570/SAP_001.pdf